CLINICAL TRIAL: NCT01997450
Title: A Case Control Study of the Effectiveness of Q/LAIV Versus Inactivated Influenza Vaccine and No Vaccine in Subjects 2-17 Years of Age
Acronym: ICICLE
Status: Terminated | Type: Observational
Why Stopped: FDA did not require the fourth season of recruitment as planned originally. Study closed.
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-VA-MEDI3250-1116
Record Dates: First submitted 2013-11-06; First posted 2013-11-28 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Influenza Vaccine Effectiveness
Keywords: Q/LAIV/FluMist® Quadrivalent Vaccine; Inactivated Influenza Vaccine (IIV); Effectiveness; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A nasal swab specimen will be collected and tested for influenza and other viral pathogens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Q/LAIV: FluMist Quadrivalent
- Inactivated Influenza Vaccine: Inactivated Influenza Vaccine

SUMMARY:
This is a post-marketing case-controlled study of the effectiveness of a quadrivalent live attenuated influenza vaccine (Q/LAIV/FluMist® Quadrivalent) versus Inactivated Influenza Vaccine (IIV) and No Vaccine in subjects 2-17 years of age.

DETAILED DESCRIPTION:
This post-marketing study will enroll approximately 5,200 subjects 2-17 years of age who are seeking care in an outpatient setting for febrile acute respiratory illness. This study will begin in the fall of 2013 and will be completed after 4 influenza seasons (i.e.after the 2016-2017 influenza season). No investigational product will be administered in this study. A nasal swab will be obtained and tested for the presence of influenza virus and other viral pathogens. This study will be conducted at 4 sites in the United States of America. The duration of study participation for each subject is one day.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling children and adolescents 2 to 17 years of age.
* Written Informed Consent or Assent.
* Acute respiratory illness documented at study visit or at home with fever (oral temperature ≥ 100.0° Fahrenheit at study visit, or history of fever reported by parents, or use of antipyretic prior to study visit)
* Symptom onset less than 5 days prior to study visit.
* Subject and/or subject's legal representative is able to understand and comply with the requirements of the protocol as judged by the investigator.

Exclusion Criteria:

* Treatment with an antiviral drug for influenza (oseltamivir or Tamiflu®, zanamivir or Relenza®) during the 14 days before enrollment
* Any condition that, in the opinion of the investigator, would interfere with interpretation of subject safety or study results
* Concurrent enrollment in another clinical study

Patient already enrolled during this influenza season

* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects 2 to 17 years of age who are seeking care in an outpatient setting for febrile acute respiratory illness.
Sampling Method: Non-Probability Sample
Enrollment: 4121 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Identification of cases positive for wild-type influenza with an end-point PCR genotyping assay. | Up to 6 months for each individual flu season
  Vaccine Effectiveness is defined as 100 x (1-odds ratio), where the odds ratio is the odds of exposures (Q/LAIV versus Inactivated Influenza Vaccine or no vaccine) among laboratory confirmed cases of flu versus controls. Effectiveness will be monitored by flu season, class of age and by influenza strain.

CONTACTS AND LOCATIONS:
Overall Officials: Herve Caspard, MD, Study Director — MedImmune LLC
Locations (12):
- United States (8):
  - Research Site, Gainesville, Florida
  - Research Site, Bloomington, Minnesota
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, Temple, Texas
  - Research Site, Marshfield, Wisconsin
- United Kingdom (4):
  - Research Site, Bristol
  - Research Site, Oxford
  - Research Site, Southampton
  - Research Site, Tooting

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Poehling KA, Caspard H, Peters TR, Belongia EA, Congeni B, Gaglani M, Griffin MR, Irving SA, Kavathekar PK, McLean HQ, Naleway AL, Ryan K, Talbot HK, Ambrose CS. 2015-2016 Vaccine Effectiveness of Live Attenuated and Inactivated Influenza Vaccines in Children in the United States. Clin Infect Dis. 2018 Feb 10;66(5):665-672. doi: 10.1093/cid/cix869. PMID 29029064
- [Derived] McLean HQ, Caspard H, Griffin MR, Poehling KA, Gaglani M, Belongia EA, Talbot HK, Peters TR, Murthy K, Ambrose CS. Effectiveness of live attenuated influenza vaccine and inactivated influenza vaccine in children during the 2014-2015 season. Vaccine. 2017 May 9;35(20):2685-2693. doi: 10.1016/j.vaccine.2017.03.085. Epub 2017 Apr 10. PMID 28408121
- [Derived] Caspard H, Coelingh KL, Mallory RM, Ambrose CS. Association of vaccine handling conditions with effectiveness of live attenuated influenza vaccine against H1N1pdm09 viruses in the United States. Vaccine. 2016 Sep 30;34(42):5066-5072. doi: 10.1016/j.vaccine.2016.08.079. Epub 2016 Sep 6. PMID 27613072
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=MA-VA-MEDI3250-1116&attachmentIdentifier=e0d0f524-6632-4915-9806-fd62d9703860&fileName=Redacted_CSR_Synopsis.pdf&versionIdentifier=